CLINICAL TRIAL: NCT02108678
Title: One-Day Intervention for Depression and Impairment in Migraine Patients
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Lilian Dindo, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201301712
Record Dates: First submitted 2014-03-28; First posted 2014-04-09 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Migraine; Depression
Keywords: Acceptance and Commitment Therapy (ACT); Depression; Illness Management; Behavioral Treatment; Impairment
MeSH Terms: conditions — Migraine Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-ME (Experimental): ACT-ME is designed to reduce behavioral avoidance and to enhance acceptance-based coping. It includes: 1) Behavioral Change Training involving a) teaching patients how to recognize ineffective patterns of behavior and habits, b) exploring and setting life goals and goals related to mental and physical health, and c) promoting effective and committed actions to achieve these goals despite the urge to do otherwise; 2) Acceptance and Mindfulness Training emphasizing new ways of managing troubling thoughts, feelings, and physical sensations; and 3) Migraine education whereby each of the educational topics listed below will be covered without detailed discussion of the topics.
  Interventions: Behavioral: ACT-ME
- Migraine Education Only (Experimental): The MEO workshop will last six hours and involve educating participants about migraine, its natural course, its prodromal symptoms and triggers for symptom worsening, risk for migraine chronification, how to use abortive migraine medications, medication overuse headache, medical and psychological treatments of migraine, migraine comorbidity, and menstrual migraine. The group leaders will present one educational topic at a time and the participants will discuss and reflect about issues and experiences related to the topic. If necessary, the group leaders will raise specific discussion questions to facilitate group dialogue and participant involvement. However, information on coping practices will be omitted.
  Interventions: Behavioral: Migraine Education Only

INTERVENTIONS:
Behavioral: ACT-ME — 1 hour discussion about migraine education (ME) and 5 hours of group therapy based on Acceptance and Commitment Therapy (ACT). Migraine education covers topics including migraine symptoms, triggers for worsening of migraine symptoms, how to use migraine medications, medication overuse headache, etc. The ACT intervention includes: 1) Behavioral Change Training and; 2) Mindfulness and Acceptance Training emphasizing new ways of managing troubling thoughts, feelings, and physical sensations.
  Other Names: Acceptance and Commitment Training Plus Migraine Education
  Arms: ACT-ME
Behavioral: Migraine Education Only — 6 hour discussion of migraine education only (MEO). This will involve educating participants about migraine, its natural course, its prodromal symptoms and triggers for symptom worsening, risk for migraine chronification, how to use abortive migraine medications, medication overuse headache, medical and psychological treatments of migraine, migraine comorbidity, and menstrual migraine.
  Other Names: Illness Management
  Arms: Migraine Education Only

SUMMARY:
The purpose of this research study is to examine whether a one-day group workshop, integrating principles from Acceptance and Commitment Therapy and Migraine Education, will result in greater improvements in depressive symptoms and functioning impairment in patients with comorbid migraine and depression than a similar one-day group workshop with Migraine Education only.

DETAILED DESCRIPTION:
Adults with comorbid depression and migraine will be randomized to a 1-day (6-hour) workshop of Acceptance and Commitment Training + Migraine Education (ACT-ME) or Migraine Education only (MEO). The intervention delivered to both study arms will be identical except for the addition of the ACT component delivered in the ACT-ME condition, thereby allowing an estimate of the specific additive effect of the psychotherapy. Measures of acceptance and behavioral avoidance, theoretically important mechanisms of change, will be used to test intervention components by examining whether these processes are uniquely affected by the ACT-ME intervention and whether they account for observed treatment effects. The central hypothesis is that the ACT-ME treatment will lead to significantly greater reduction in depression (HRSD) and disability (WHO-DAS, WHOQOL, and HDI) at follow-up compared to the MEO treatment. ACT-ME participants also are expected to demonstrate reductions in behavioral avoidance and enhanced acceptance, which mediate treatment effects. Treatment gains are expected to be maintained through the 6-month follow-up.

Aim 1: To examine the efficacy of a 1-day ACT-ME intervention compared to MEO for treating depression in patients with comorbid depression and migraine.

Hypothesis 1: At 3- and 6-month follow-up, ACT-ME will be more efficacious than MEO as assessed by: 1) a significantly greater decline on the Hamilton Rating Scale for Depression (HRSD) total score; 2) a significantly higher proportion of participants showing 50% or greater decline on the HRSD; and 3) a significantly higher proportion of participants no longer meeting depression criteria on SCID-IV.

Aim 2: To examine the efficacy of a 1-day ACT-ME intervention compared to MEO on functioning in patients with comorbid depression and migraine.

Hypothesis 2: At 3- and 6-month follow-up, compared to the MEO group, participants in the ACT-ME group will exhibit significantly greater improvement in functioning (measured by World Health Organization Disability Assessment Schedule-Total Score; WHO-DAS) and quality of life (measured by World Health Organization Quality of Life Total; WHO-QOL), and greater decline in headache-related disability (measured by Headache Disability Inventory; HDI).

Aim 3: To determine whether changes in acceptance-based coping and behavioral avoidance will mediate the changes in depressive symptoms and disability.

Hypothesis 3: Increases in acceptance-based coping and reductions in behavioral avoidance will mediate relations between treatment group and 1) decline in depressive symptoms as measured by the HRSD and 2) disability, as measured by the WHO-DAS and HDI. Acceptance and Behavioral Avoidance will be measured using the Acceptance and Action Questionnaire and Chronic Pain Acceptance Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-65
* Current major depressive episode on the SCID-IV (46)
* Score of ≥ 17 on the HRSD (47)
* Confirmation of diagnosis of migraine from medical record
* 4-12 migraines in the previous month

Exclusion Criteria:

* Bipolar, psychotic, or current substance use disorders
* History of brain injury
* Imminent suicidality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
HRSD | 24 weeks
  The HRSD is a structured clinical interview for depression severity. Change from baseline measured at 2, 6, 12, and 24 weeks post workshop.
SCID-IV | 24 weeks
  Semi-structured clinical interview for depression. Change from baseline measured at 12 and 24 weeks post workshop.

SECONDARY OUTCOMES:
WHO-DAS-II | 24 weeks
  This is a self-report questionnaire that measures difficulties due to physical and mental health conditions. Measure change from baseline at 12 and 24 weeks post-workshop.
WHO-QOL | 24 weeks
  The WHO-QOL is a self-report measure that assesses four domains of quality of life: physical health, psychological well-being, social relationships, and environment. Measure change from baseline at 12 and 24 weeks post workshop.
HDI | 24 weeks
  The HDI is a self-report measure that assesses the burden of headaches through perceived impact of headaches on functioning. Measure changes from baseline at 12 and 24 weeks post workshop.

OTHER OUTCOMES:
AAQ-II | 24 weeks
  The AAQ-II is a self-report measure that assesses experiential avoidance, or the tendency to avoid unwanted internal experiences (e.g., "I try hard to avoid feeling depressed or anxious"), as well as acceptance, the term used to describe the counter process (e.g., "My thoughts and feelings do not get in the way of how I want to live my life"). Measure changes from baseline at 2, 6, 12, and 24 weeks post workshop.
CPAQ | 24 weeks
  The CPAQ is a self-report measure that assesses Activity Engagement, the degree to which one engages in life activities regardless of pain, and Pain Willingness, the willingness to have pain without trying to avoid or reduce it. Measure change from baseline at 2, 6, 12, and 24 weeks post workshop.
Demographics Questionnaire | 1 day
  The following information will be obtained: age, ethnicity, marital status, educational level, household income, occupation, current mental health treatment, current medication, number of migraines in previous month, and age of onset of migraine. Information will only be obtained at initial meeting.
Treatment Questionnaire | 24 weeks
  Changes in medications and involvement in psychotherapy/counseling will be documented at each contact and will be confirmed by reviewing medical and pharmacy records. Measured at baseline and 2, 6, 12, and 24 weeks post workshop.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Carver College of Medicine Department of Psychiatry, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Dindo LN, Recober A, Calarge CA, Zimmerman BM, Weinrib A, Marchman JN, Turvey C. One-Day Acceptance and Commitment Therapy Compared to Support for Depressed Migraine Patients: a Randomized Clinical Trial. Neurotherapeutics. 2020 Apr;17(2):743-753. doi: 10.1007/s13311-019-00818-0. PMID 31863406